CLINICAL TRIAL: NCT03284242
Title: Tolerance Induction Using Autologous Regulatory T Cell Infusion and Zortress (Everolimus) in Renal Transplant Recipients: a Pilot Study
Brief Title: A Pilot Study Using Autologous Regulatory T Cell Infusion Zortress (Everolimus) in Renal Transplant Recipients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Roberto Gedaly (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Roberto Gedaly, Sponsor/Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-0779-F6A; CRAD001AUS210T (Other Grant/Funding Number: Novartis)
Record Dates: First submitted 2017-08-08; First posted 2017-09-15 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: End Stage Renal Disease; Kidney Transplant
Keywords: Kidney; Transplant
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Single intravenous infusion of autologous, ex vivo, expanded Treg cells in renal transplant recipients who are on Everolimus-based immunosupressive therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous Treg Infusion (Experimental): This will be a single intravenous (IV) infusion. A participant's own expanded regulatory T cells will be added to Albumin, and administered to them. The amount of the solution will be approximately 300 ml and the infusion will take about 3 to 4 hours.
  Interventions: Drug: Treg

INTERVENTIONS:
Drug: Treg — Collect white blood cells to isolate Treg cells for expansion. Once the blood cells are collected the cells will be cultured in the laboratory and will be expanded. After approximately 3 weeks in culture, the cells will have increased in number and be ready for the autologous Treg cell infusion.
  Other Names: regulatory T cells

SUMMARY:
This study will enroll individuals who have end stage renal disease and who are undergoing a solitary kidney transplant. This study is investigating/evaluating the safety and effectiveness of collecting, expanding and infusing a specific certain type of immune cell known as Regulatory T cells (Treg cells) to renal transplant recipients who are using Zortress (Everolimus) as immunosuppressive therapy.

Treg cells, once they have been expanded in the laboratory to help prevent kidney rejection. Treg cells are collected from a participant's blood through a procedure called apheresis. Treg cells are a type of white blood cells that are able to suppress the activity of other immune cells responsible for organ rejection. The investigator plans to enroll 12 participants at the University of Kentucky.

DETAILED DESCRIPTION:
The purpose of this research study is to learn alternative ways to control the body's immune responses after renal transplantation. The investigator's goal is to prevent or reduce the side-effects of long-term immunosuppressive therapy.

By doing this study, the investigator hopes to learn how safe and effective infusing autologous Treg cells, after renal transplantation, to renal transplant recipients who are taking Zortress (Everolimus) to control the immune response.

Individuals who decide to take part in this research study and are eligible to start, will be followed for 1 year after their transplant. The research procedures will be conducted at the University of Kentucky Medical Center and require nine study visits. One of the study visits requires an overnight stay. Participants will be admitted to the University of Kentucky Center for Clinical and Translational Science (CCTS) inpatient research unit for this study visit. Depending on the frequency of an participant's post-transplant clinic visits, some of the study visits could be done at the same time as their regular clinic visits. If not, they will occur in the transplant clinic or in the University of Kentucky Center for Clinical and Translational Science (CCTS) outpatient research unit.

The total amount of time required for participation in the study will be up to 40 hours over 1 year. The total amount of blood taken for the study will be about 14 tablespoons (200ml/6.5 ounces) over 1 year.

STUDY PROCEDURES:

Blood Samples: These will be collected via a needle inserted into a vein in the arm.

Human immunodeficiency virus (HIV) and hepatitis testing: Test for HIV, Hepatitis B and Hepatitis C will be done as part of the participant's routine transplant evaluation. The results from these tests will be used to determine study eligibility at the pre-transplant study visit.

If any of these tests are positive, a qualified person will provide counseling to the participant. The State of Kentucky requires that researchers must report HIV, Hepatitis B and Hepatitis C positive test results to the local health department serving the jurisdiction in which the participant resides, and that the information reported must include the participant's full name, address, phone number, county of residence, and applicable disease/condition.

Apheresis: Apheresis is a procedure in which a machine receives blood removed from a participant's body and separates it into its various components: plasma, platelets, white blood cells and red blood cells. This procedure is done in the Apheresis Center in the Gill Heart Building at the UK Chandler Hospital. Depending on the reason for apheresis, one of these components is isolated and collected by the instrument, while the others are re-infused to the body.

In this particular research study the investigator is going to collect white blood cells to isolate Treg cells for expansion. The process of collecting white blood cells will take approximately 90 minutes. Once the blood cells are collected, the research team will isolate the Treg cells. These cells will be cultured in the laboratory under special conditions and will be expanded. After approximately 3 weeks in culture, the cells will have increased in number and be ready for the autologous Treg cell infusion.

Autologous Treg cell infusion: This will be a single intravenous (IV) infusion. A standard IV line will be started in a vein of the arm. The participant's own expanded regulatory T cells will be added to a sterile infusion solution, called Albumin, and administered to to the participant, and the infusion will take about 3 to 4 hours. Participant's vital signs will be monitored before, during, and after the infusion.

Renal Biopsy: Two renal biopsies (removal of a piece of kidney tissue) will be performed. The first one will be done in the operating room during the participant's renal transplant surgery. The biopsy will come from the new kidney prior to being transplanted. The second one will be done 6 weeks after the autologous Treg cell infusion and will be compared to the first one. The second renal biopsy is optional. If a participant agrees to the second biopsy it will be done as an outpatient procedure in the radiology department at the University of Kentucky. Using an ultrasound for guidance, the investigator will pass a larger needle through the skin to obtain a small sample of the transplanted kidney.

Physical Examination and Vital Sign Measurement: These will be done by a member of the study team. The participant's body temperature, heart rate, respiratory rate, and blood pressure will be measured and recorded.

Pregnancy Tests: A pregnancy test will be performed on women who could be pregnant prior to beginning the study and again prior to receiving the autologous Treg cell infusion to exclude the possibility of pregnancy. For study purposes women who could become pregnant must use two effective contraceptive starting prior to renal transplant through to visit 9.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English able to understand and provide informed consent
* End stage renal disease listed for primary solitary kidney transplant
* Willing to participate in the study and comply with study requirements
* Female participants must agree to use 2 different birth control methods

Exclusion Criteria:

* History of previous organ, tissue or cell transplant
* Known sensitivity to Sirolimus, Everolimus, Tacrolimus or MMF
* Previous chronic use of systemic glucocorticoids or other immunosuppression, or biologic immunomodulators
* Significant or active infection: HIV, Hepatitis B and C
* Active cancer or history of cancer within 3 years of screening
* Participation in other study that involved investigational drug or regimens in the preceding 12 months
* History of delayed or abnormal wound healing
* Delayed graft function
* Chronic illness or prior treatment which, in the opinion of the investigator, precludes study participation
* Pregnant or breastfeeding or refusal to us birth control
* Inability or unwillingness to comply with study protocol or procedures
* Chronic use of anticoagulants
* Blood transfusion 3 months prior to transplant
* History of non-compliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Changes in Tregs Infusion Toxicities | Immediately following Tregs infusion and again within 24 hours after Tregs infusion
  Laboratory measurement and observed toxicities immediately and with in 24 hours post infusion of Tregs.
Changes in Kidney Function | for 2 years from the start of the study
  Creatinine level measurement
Changes In Steroid Resistance Rejection Rates | 1, 6 and 12 months post Tregs infusion
  Laboratory measurement
Infectious Complications | for 2 years from the start of the study
  Laboratory measurement

SECONDARY OUTCOMES:
Treg cell measurements within the allograft | 6 to 12 weeks post transplant
  Renal biopsy
Circulating T cell subset measurements | twice a week for 4 weeks then weekly for 3 months
  laboratory analysis

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Gedaly, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gedaly R, De Stefano F, Turcios L, Hill M, Hidalgo G, Mitov MI, Alstott MC, Butterfield DA, Mitchell HC, Hart J, Al-Attar A, Jennings CD, Marti F. mTOR Inhibitor Everolimus in Regulatory T Cell Expansion for Clinical Application in Transplantation. Transplantation. 2019 Apr;103(4):705-715. doi: 10.1097/TP.0000000000002495. PMID 30451741